CLINICAL TRIAL: NCT01301755
Title: Diagnosis of Invasive Pulmonary Aspergillosis by Direct Lung Tissue Aspergillus Galactomannan Antigen Detection From Aspirate by Ultrasound-guided Fine Needle Aspiration
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Hao-Chien Wang, Medical department of National Taiwan University Hospital
Other Study IDs: 201002035R
Record Dates: First submitted 2010-03-17; First posted 2011-02-23 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Immunocompromised

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Procedure: Lung aspiration

INTERVENTIONS:
Procedure: Lung aspiration — direct lung tissue Aspergillus galactomannan antigen detection from aspirate by ultrasound-guided fine needle aspiration

SUMMARY:
Invasive aspergillosis is a serious and often fatal infection in patients who are neutropenic or have undergone solid organ or stem cell transplantation. However, early diagnosis of invasive aspergillosis is a challenge. Reiss and Lehmann first described the value of serum Galactomanna (GM) for diagnosis of invasive pulmonary aspergillosis in 1979. The availability of the Platelia Aspergillus, a sandwich ELISA that has been approved by FDA in 2003 for managing patients at risk of invasive aspergillosis because of the early detection of the GM antigen. In several studies so far the specificity of the serum galactomannan assay was greater than 85%; however, variable sensitivity from 29~100% was noted over years. In addition, low values and false-negative results are seen more often in nonneutropenic and solid organ transplantation patients as opposed to severely granulocytopenic patients .There are several factors that might explain the reported difference in the performance of antigen detection, including the biological factors and epidemiological factors.

In recent years, specimens of other body fluids are increasingly used for detection of Aspergillus galactomannan antigen, including urine, bronchoalveolar lavage(BAL) fluid, cerebrospinal fluid and even the tissue specimen. However, the sensitivity and specificity of the GM detection in various specimens still have considerably variation. Ultrasound-guided transthoracic aspirate is a safe and useful method for collecting specimens for accurate bacteriologic diagnosis of lung abscess and obstructive pneumonitis10. We also reported a study of diagnosis of pulmonary Cryptococosis by ultrasound guided percutaneous aspiration. We plan to perform a prospective single-center study to investigate the role of GM in the target organ (lung tissue/fluid) by using ultrasound-guided fine needle aspirate for early diagnosis invasive aspergillosis compared with the serum galactomannan.

DETAILED DESCRIPTION:
Invasive aspergillosis is a serious and often fatal infection in patients who are neutropenic or have undergone solid organ or stem cell transplantation. However, early diagnosis of invasive aspergillosis is a challenge. Reiss and Lehmann first described the value of serum Galactomanna (GM) for diagnosis of invasive pulmonary aspergillosis in 1979. Galactomannan is a water-soluble, polysaccharide cell wall component which is released by Aspergillus during fungal growth after inhalation of Aspergillus conidia to the lung. The availability of the Platelia Aspergillus, a sandwich ELISA that has been approved by FDA in 2003 for managing patients at risk of invasive aspergillosis because of the early detection of the GM antigen. In several studies so far the specificity of the serum galactomannan assay was greater than 85%; however, variable sensitivity from 29~100% was noted over years. In addition, low values and false-negative results are seen more often in nonneutropenic and solid organ transplantation patients as opposed to severely granulocytopenic patients .There are several factors that might explain the reported difference in the performance of antigen detection, including the biological factors (non-neutropenic patients, prior exposure to antifungal agents, encapsulation abscess preventing GM leakage to the circulation, renal clearance,…etc.) and epidemiological factors (patient population, cut-off value, prevalence of infection…etc) .

In recent years, specimens of other body fluids are increasingly used for detection of Aspergillus galactomannan antigen, including urine, bronchoalveolar lavage(BAL) fluid, cerebrospinal fluid and even the tissue specimen. However, the sensitivity and specificity of the GM detection in various specimens still have considerably variation. Ultrasound-guided transthoracic aspirate is a safe and useful method for collecting specimens for accurate bacteriologic diagnosis of lung abscess and obstructive pneumonitis10. We also reported a study of diagnosis of pulmonary Cryptococosis by ultrasound guided percutaneous aspiration. We plan to perform a prospective single-center study to investigate the role of GM in the target organ (lung tissue/fluid) by using ultrasound-guided fine needle aspirate for early diagnosis invasive aspergillosis compared with the serum galactomannan.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients with following host factors:

* A hematologic malignancy, unless they were already treated with antifungals for a presumed or proven IA
* Cancer and receiving chemotherapy within the last 3 months before admission
* Solid organ transplant recipient
* Prolong steroid use
* Recipient of any other immunosuppressive treatment (tacrolimus, cyclosporine, methotrexate, cyclophosphamide, sirolimus)
* Child C cirrhosis
* HIV
* Febrile neutropenia

Combined at least two of the three following features:

* Fever(>37.5。C) refractory to at least 3 days of appropriate antibiotics or Fever relapsing after a period of defervescence of at least 48 hours while still receiving antibiotics
* Clinical signs and/or symptoms suggestive of invasive mycosis: pleuritic chest pain or physical finding of pleural rub, or one of the following symptoms of lower respiratory tract infection (new sputum secretions, dypsnea, or hemoptysis)
* Development of new pulmonary infiltrates on chest X-ray or HRCT

Exclusion Criteria:

* Patients who can't be cooperative
* Have bleeding tendency or coagulopathy (PLT<100K)
* Pulmonary lesion could not identify by chest ultrasonography
* Patients who do not have informed consent before the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: immunocompromised patients
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
The diagnostic rate of lung tissue Aspergillus galactomannan antigen detection compaired with serum Aspergillus galactomannan antigen detection | 3 weeks
  we will use echo-guide lung tissue aspiration to detect lung tissue Aspergillus galactomannan antigen compaired with conventional serum Aspergillus galactomannan antigen detection to early diagnose pulmonary aspergillosis

CONTACTS AND LOCATIONS:
Overall Officials: Hao-Chien Wang, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan